CLINICAL TRIAL: NCT03687450
Title: Feasibility of a Yoga- and Mindfulness-Based Intervention for Resident Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Kripalu Center for Yoga and Health (Other)
Responsible Party: Principal Investigator, Sat Bir Khalsa, PhD, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P002372
Record Dates: First submitted 2018-03-27; First posted 2018-09-27 (Actual); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Burnout, Professional; Anxiety; Depression; Stress
Keywords: yoga; mindfulness; meditation; resident; residency
MeSH Terms: conditions — Burnout, Professional; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Yoga) Arm (Experimental): Received a weekly 60-minute yoga-based class over 6 weeks with direction for a 5-10 minute daily home practice.
  Interventions: Behavioral: RISE yoga-based program
- No-treatment Control Arm (No Intervention): Waitlist control-- group received one session of yoga-based class at the completion of the study.

INTERVENTIONS:
Behavioral: RISE yoga-based program — The RISE program developed by Kripalu Center for Yoga and Health includes yoga postures, mindfulness practices, meditation, breathing techniques, and education sessions about mindful approaches to daily living. The RISE program will be delivered as a 6-week yoga-based program on-site at Brigham and Women's Hospital in Boston, MA. The program will consist of six 60-90-minute weekly yoga-based RISE classes. Sessions will be lead by experienced instructors from Kripalu Center for Yoga & Health. Subjects in this arm will also be asked to participate in 5-10 minutes of daily home practice with direction from the RISE curriculum.
  Arms: Intervention (Yoga) Arm

SUMMARY:
The investigators aim to initiate and complete the first investigation of the effect of a yoga-based program on resident physicians' psychological health using a randomized controlled trial to assess feasibility of the program in this population and measure outcomes across several domains. To meet the goals of the proposed project the investigators have identified 3 specific aims:

Specific Aim 1: Assess the acceptability and feasibility of the yoga program through measuring participation and conducting standardized interviews with a subset of yoga participants.

Specific Aim 2: Evaluate the effect of the yoga program on resident physicians' stress, burnout, resilience, mindfulness, mood, depression, anxiety, and sleep quality using quantitative self-report measures.

Specific Aim 3. Examine whether outcome measures were perceived as relevant to the participants' work environment and were not burdensome as to the length and content of the program.

DETAILED DESCRIPTION:
The project will implement a single group mixed-methods randomized controlled trial to investigate the impact of the 6-week RISE program on psychological health in Longwood medical area residents. The RISE program is an existing standardized yoga program at Kripalu that will be adapted for residents in a 60-90-minute, once-weekly class for six weeks. Participants will be randomized to either the RISE yoga program or a no-treatment control group. Participants randomized to the RISE program will also be instructed to maintain a short 10-15-minute daily home yoga practice. Sessions will be lead by experienced instructors from Kripalu and will be held in the Longwood medical area. Self-report outcomes will be assessed at baseline, at program completion (post-program), at 2-month follow-up, and at 6-month follow-up.

Participants will include resident physicians at Longwood medical area hospitals. The only exclusion criterion is having practiced yoga, meditation, tai chi, qigong, or another mind-body practice at least 25 hours or more in the past 6 months. Participants must be willing not to practice mind-body programs other than the treatment protocol during the intervention. We plan to enroll up to 200 participants with a goal of at least 60 participants with a 2:1 ratio of participants randomized to yoga to participants randomized to control. The control group will receive one session of RISE after their participation in the trial is complete.

ELIGIBILITY:
Inclusion Criteria:

* Individuals enrolled in residency programs at Brigham and Women's Hospital, Beth Israel Deaconess, Boston Children's Hospital, or a Harvard Combined Residency Program
* Individuals must be willing to not practice mind-body programs other than the intervention during the treatment protocol
* Must be proficient in English

Exclusion Criteria:

* Individuals who currently practice yoga, meditation, tai chi, qigong, and other mind-body practices more than 25 hours in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sat Bir Khalsa, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagnild GM, Young HM. Development and psychometric evaluation of the Resilience Scale. J Nurs Meas. 1993 Winter;1(2):165-78. PMID 7850498
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Baer RA, Carmody J, Hunsinger M. Weekly change in mindfulness and perceived stress in a mindfulness-based stress reduction program. J Clin Psychol. 2012 Jul;68(7):755-65. doi: 10.1002/jclp.21865. Epub 2012 May 23. PMID 22623334
- [Background] Gu J, Strauss C, Crane C, Barnhofer T, Karl A, Cavanagh K, Kuyken W. Examining the factor structure of the 39-item and 15-item versions of the Five Facet Mindfulness Questionnaire before and after mindfulness-based cognitive therapy for people with recurrent depression. Psychol Assess. 2016 Jul;28(7):791-802. doi: 10.1037/pas0000263. Epub 2016 Apr 14. PMID 27078186
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] West CP, Dyrbye LN, Sloan JA, Shanafelt TD. Single item measures of emotional exhaustion and depersonalization are useful for assessing burnout in medical professionals. J Gen Intern Med. 2009 Dec;24(12):1318-21. doi: 10.1007/s11606-009-1129-z. Epub 2009 Oct 3. PMID 19802645
- [Background] West CP, Dyrbye LN, Satele DV, Sloan JA, Shanafelt TD. Concurrent validity of single-item measures of emotional exhaustion and depersonalization in burnout assessment. J Gen Intern Med. 2012 Nov;27(11):1445-52. doi: 10.1007/s11606-012-2015-7. Epub 2012 Feb 24. PMID 22362127
- [Background] Trockel M, Bohman B, Lesure E, Hamidi MS, Welle D, Roberts L, Shanafelt T. A Brief Instrument to Assess Both Burnout and Professional Fulfillment in Physicians: Reliability and Validity, Including Correlation with Self-Reported Medical Errors, in a Sample of Resident and Practicing Physicians. Acad Psychiatry. 2018 Feb;42(1):11-24. doi: 10.1007/s40596-017-0849-3. Epub 2017 Dec 1. PMID 29196982
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Pilkonis PA, Yu L, Dodds NE, Johnston KL, Maihoefer CC, Lawrence SM. Validation of the depression item bank from the Patient-Reported Outcomes Measurement Information System (PROMIS) in a three-month observational study. J Psychiatr Res. 2014 Sep;56:112-9. doi: 10.1016/j.jpsychires.2014.05.010. Epub 2014 May 29. PMID 24931848
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Dyrbye LN, Satele D, Sloan J, Shanafelt TD. Ability of the physician well-being index to identify residents in distress. J Grad Med Educ. 2014 Mar;6(1):78-84. doi: 10.4300/JGME-D-13-00117.1. PMID 24701315

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention (Yoga) Arm: This is the group that will receive a weekly 60-90minute yoga-based class for six weeks and direction for a 5-10 minute daily home practice.
  RISE yoga-based program: The RISE program developed by Kripalu Center for Yoga and Health includes yoga postures, mindfulness practices, meditation, breathing techniques, and education sessions about mindful approaches to daily living. The RISE program will be delivered as a 6-week yoga-based program on-site at Brigham and Women's Hospital in Boston, MA. The program will consist of six 60-90-minute weekly yoga-based RISE classes. Sessions will be lead by experienced instructors from Kripalu Center for Yoga & Health. Subjects in this arm will also be asked to participate in 5-10 minutes of daily home practice with direction from the RISE curriculum.
- No-treatment Control Arm: This group will receive no intervention during the study. At the conclusion of the study, this group will receive one free yoga-based class.
Period: Overall Study
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Started | 38 | 18
Post-Program Follow-Up | 28 (1 withdrew, 9 lost to follow-up) | 15 (3 lost to follow-up)
Two-month Follow-up | 26 (2 lost to follow-up) | 16 (2 lost to follow-up (N.B. 1 participant completed 2-month follow-up but not post-program follow-up))
Completed | 26 | 16
Not Completed | 12 | 2

BASELINE CHARACTERISTICS:
Population: Participants included in analysis were those who completed ANY follow-up survey (post-program or two-month follow-up). This includes 28 who completed post-program follow-up in intervention arm and 16 who completed two-month follow-up in control arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm | Total
Number analyzed (Participants) | 28 | 16 | 44
Age, Continuous [Mean (Full Range); unit: years] | 29.3 [26 to 33] | 29.1 [27 to 33] | 29.2 [26 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 26 | 14 | 40
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 10 | 28
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 0 | 1
Year in Training [Count of Participants; unit: Participants]
  1st year | 9 | 3 | 12
  2nd year | 6 | 5 | 11
  3rd year | 8 | 3 | 11
  4th year and above | 5 | 5 | 10
Specialty [Count of Participants; unit: Participants]
  Internal Medicine | 12 | 8 | 20
  OB/GYN | 3 | 2 | 5
  Diagnostic Radiology | 3 | 2 | 5
  Emergency Medicine | 2 | 0 | 2
  Psychiatry | 4 | 2 | 6
  Medicine-Pediatrics | 1 | 0 | 1
  Anesthesiology | 3 | 1 | 4
  Physical Medicine & Rehabilitation | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Attending the Yoga Program
Description: Participants were ask to rate the feasibility of attending the yoga program on a visual analogue scale from 0 (not at all feasible) to 100 (very feasible). Only the intervention group rated feasibility since the control group was a waitlist control group and did not attend the program. The standard deviation of the mean score was calculated.
Time Frame: Post-program
Population: Participants analyzed included those in the intervention group who completed any follow-up timepoint, including post-program and/or two-month follow-up. Since the waitlist control group did not attend the program, they were not asked to assess feasibility.
Measure: Mean (Standard Deviation); unit: visual analogue scale, 0 to 100
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Number analyzed (Participants) | 28 | 0
visual analogue scale, 0 to 100 | 28.9 (25.6) |

2. Secondary Outcome: Difference in Burnout
Description: Maslach Burnout Inventory (short form, 2 items) - scores from 0-12; higher is more burnout
Time Frame: Post-program and 2-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Number analyzed (Participants) | 28 | 16
score on a scale
  Baseline | 6.23 (0.52) | 6.33 (0.92)
  Post-program | 5.65 (0.50) | 6.83 (0.66)
  2-month follow-up | 5.72 (0.53) | 6.43 (0.99)

3. Secondary Outcome: Difference in Professional Fulfillment
Description: Professional Fulfillment Index (PFI; 16 items) - scores from 0-4 for professional fulfillment scale; higher is more fulfillment
Time Frame: Baseline, post-program, and 2-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Number analyzed (Participants) | 28 | 16
score on a scale
  Baseline | 1.70 (0.12) | 1.53 (0.18)
  Post-program | 1.35 (0.14) | 1.48 (0.20)
  2-month follow-up | 1.38 (0.10) | 1.56 (0.21)

4. Secondary Outcome: Difference in Resident Well-being
Description: Resident Well-Being Index (7 items) - scores from 0-7; higher is worse wellbeing
Time Frame: Baseline, post-program, and 2-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Number analyzed (Participants) | 28 | 16
score on a scale
  Baseline | 4.19 (0.30) | 4.08 (0.58)
  Post-program | 3.15 (0.33) | 3.62 (0.35)
  2-month follow-up | 3.40 (0.37) | 3.25 (0.49)

5. Secondary Outcome: Difference in Resilience
Description: Resilience Scale (RS-14; 14 items) - scores from 14-98; higher more resilience
Time Frame: Baseline, post-program, and 2-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Number analyzed (Participants) | 28 | 15
score on a scale
  Baseline | 70.61 (2.26) | 71.20 (3.14)
  Post-program | 76.32 (1.79) | 72.07 (3.02)
  2-month follow-up | 72.61 (1.76) | 72.43 (3.22)

6. Secondary Outcome: Difference in Mindfulness
Description: Five Facet Mindfulness Questionnaire (FFMQ; short form, 15 items) - scores from 15-75; higher score means more mindfulness
Time Frame: Baseline, post-program, and 2-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Number analyzed (Participants) | 28 | 16
score on a scale
  Baseline | 48.54 (1.14) | 48.60 (1.92)
  Post-program | 54.27 (1.42) | 49.73 (1.54)
  2-month follow-up | 51.83 (0.99) | 48.56 (1.49)

7. Secondary Outcome: Difference in Stress
Description: Perceived Stress Scale (PSS; 10 items) - scores from 0-40; higher is more stress
Time Frame: Baseline, post-program, and 2-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Number analyzed (Participants) | 28 | 16
score on a scale
  Baseline | 19.74 (1.09) | 20.69 (1.88)
  Post-program | 16.15 (1.38) | 18.23 (1.36)
  2-month follow-up | 16.52 (0.85) | 18.88 (1.90)

8. Secondary Outcome: Difference in Depression
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Depression (short form: depression-4) - scores from 4-20, higher is more depression
Time Frame: Baseline, post-program, and 2-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Number analyzed (Participants) | 28 | 16
score on a scale
  Baseline | 7.56 (0.64) | 7.15 (1.13)
  Post-program | 6.48 (0.54) | 7.23 (0.75)
  2-month follow-up | 7.24 (0.61) | 7.81 (0.94)

9. Secondary Outcome: Difference in Sleep Quality
Description: PROMIS Sleep Disturbance (short form, 4 items) - scores from 4-20, higher is more sleep disturbance
Time Frame: Baseline, post-program, and 2-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Number analyzed (Participants) | 28 | 16
score on a scale
  Baseline | 10.38 (0.62) | 11.62 (1.28)
  Post-program | 8.73 (0.59) | 9.92 (0.91)
  2-month follow-up | 8.96 (0.61) | 8.50 (1.02)

10. Secondary Outcome: Difference in Anxiety
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety (short form: anxiety-4) - scores from 4-20, higher is more anxiety
Time Frame: Baseline, post-program, and 2-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Number analyzed (Participants) | 28 | 16
score on a scale
  Baseline | 9.65 (0.60) | 10.00 (1.00)
  Post-program | 8.54 (0.59) | 9.15 (0.94)
  2-month follow-up | 8.96 (0.57) | 7.94 (0.81)

11. Secondary Outcome: Differences in Professional Fulfillment - Burnout Sub-Item
Description: Professional Fulfillment Index (PFI; 16 items) - scores from 0-4 for the burnout scale; higher is more burnout
Time Frame: Baseline, post-program, and 2-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
Number analyzed (Participants) | 28 | 16
score on a scale
  Baseline | 2.26 (0.13) | 1.97 (0.23)
  Post-program | 2.47 (0.15) | 2.13 (0.19)
  2-month follow-up | 2.31 (0.11) | 2.02 (0.22)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Intervention (Yoga) Arm | No-treatment Control Arm
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/18
Other Adverse Events (participants affected / at risk) | 0/38 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-05-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT03687450/Prot_000.pdf